CLINICAL TRIAL: NCT04841174
Title: The Effect of Abdominal Massage on Gastric Problems in Patients With Enteral Nutrition in Pediatric Intensive Care: A Randomized Controlled Study
Brief Title: The Effect of Abdominal Massage on Gastric Problems in Pediatric Intensive Care: A Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Sumeyye Cihan, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 202173
Record Dates: First submitted 2021-03-22; First posted 2021-04-12 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Intensive Care Units, Pediatric; Massage; Nutrition Disorders; Nurse's Role
Keywords: pediatric intensive care unit; abdominal massage; enteral nutrition; gastric problems; massage; pediatric nurse; nutrition disorders
MeSH Terms: conditions — Nutrition Disorders

STUDY DESIGN:
Intervention Model Description: The study was designed as a randomized controlled experimental study and was conducted in the pediatric intensive care unit of a training and research hospital in Istanbul between March 2021-January 2023. A total of 24 cases were included in the study, 12 in the experimental group and 12 in the control group, aged between 1 and 24 months. Randomization was performed using the urn method. Children who received mechanical ventilation support for at least 48 hours and sedation, were fully enterally fed with the same type of enteral formula, and were suitable for abdominal massage were included in the study. Abdominal massage was applied to the experimental group for 3 days, twice a day, for 15 minutes each session, while routine nursing treatment and care were provided to the control group. Abdominal circumference measurement, presence of abdominal distension, bowel sounds, vomiting and defecation frequency, and gastric residual volume amounts of the children in both groups were compared.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abdominal Massage (Experimental): Participants in the experimental group will be given an abdominal massage twice a day for 15 minutes and three days in a row by the researcher. The massage will be done 2 hours after the child has been fed. Abdominal massage will be done using the "I love u" technique.
  Interventions: Other: Abdominal massage
- Gastric measurements (No Intervention): In the experimental and control groups, the abdominal circumference will be measured by the researcher twice a day for three days in a row. The gastric residual volume will be checked during the nurses' care time. The presence of vomiting and defecation will be checked during the care time of the nurses.

INTERVENTIONS:
Other: Abdominal massage — The effect on gastric problems by applying abdominal massage to eligible participants in the study will be examined.
  Arms: Abdominal Massage

SUMMARY:
Many system functions differ in children dependent on mechanical ventilation support and may present with various complications. In the gastrointestinal system, gastric and duodenum-related decreased motility disorders are a very common problem in critically ill patients hospitalized in the intensive care unit, which increases mortality and morbidity. The prevalence of gastric dysmotility in pediatric intensive care is estimated to be 50%. Gastric problems such as vomiting, increase in the amount of gastric residue, decrease in bowel movements, abdominal distension, diarrhea/ constipation, etc. are observed as a result of the dysfunction of the gastrointestinal system. In addition to these problems; there are problems associated with the ventilator such as pneumonia, infection, bacterial growth, and stopping enteral feeding. Malnutrition as a result of stopping feeding prolongs the hospitalization of intensive care patients and affects mortality.

Intensive care nurses play a key role in providing nutritional support to patients who receive mechanical ventilation support and whose level of consciousness is reduced. Intensive care nurses have many responsibilities such as timely initiation of nutrition, application of correct nutrition, correct placement of feeding tubes, and prevention of problems that may arise as a result of nutrition. Abdominal massage practice is a therapeutic, independent, and evidence-based nursing intervention. It has been used for many years to increase the motility of the gastrointestinal system and to treat constipation. Inexpensive and easy to apply abdominal massage compared to other methods; It increases intestinal motility, accelerates the mechanical advancement of nutrients in the digestive system, improves the blood flow of the region, and is effective in reducing intra-abdominal pressure.

It has been reported in the literature that abdominal massage applied to preterm babies increases nutritional tolerance. Studies on adults have also reported that gastric residue is reduced, less vomiting is experienced, and abdominal distension is less common. However, there is no study examining the effects of abdominal massage in reducing gastrointestinal problems in children hospitalized in pediatric intensive care units and receiving ventilator support.

Therefore, the aim of this study is to examine the effect of abdominal massage on gastric problems in children who are fed enterally in the pediatric intensive care unit.

DETAILED DESCRIPTION:
According to Espen (European Society for Clinical Nutrition and Metabolism) intensive care nutrition guide; in critically ill patients under mechanical ventilation support, early enteral feeding (24-48 hours) is recommended. Nutrition, which is an important part of intensive care treatment; accelerates wound healing in critically ill patients, regulates the immune system, decreases mortality rates, and plays a role in shortening hospital stay. As a result of the early initiation of enteral feeding, the gastrointestinal system barrier mechanisms are preserved and mucosal atrophies are prevented.

Gastrointestinal, mechanical, and metabolic complications may occur in patients who are fed enterally in an intensive care unit and feeding is interrupted in these cases. Studies have shown that problems such as diarrhea, constipation, abdominal distension, aspiration pneumonia, increased gastric residual volume, and feeding intolerance occur in patients in whom enteral feeding is initiated. As a result of a study conducted with 341 children connected to mechanical ventilation, it was found that only 66.6% of the children reached their daily enteral nutrition goals on the 7th day of their hospitalization.

Massage has been used as therapeutic treatment in medicine for many years. Abdominal massage stimulates the digestive system and increases peristaltic movements. It is thought to accelerate food passage and digestion because it causes mechanical and reflexive movements in the intestines. In adult age group studies where, abdominal massage is applied; It has been reported that there is less aspiration pneumonia, the gastric residue is reduced, less vomiting is experienced and abdominal distension is less common. Similar results are seen in studies with preterm babies. It has been reported that gastric residual volume decreases, the frequency of defecation increases, and less vomiting is observed in preterm babies who are massaged. In a meta-analysis study by Biarag and Mirghafourvand, it was reported that abdominal massage reduced the frequency of vomiting and less gastric residue was removed in preterm babies. In the study conducted by Kim, it is seen that preterm babies who were massaged started enteral feeding before. In addition, it has been reported that massage helps weight gain in preterms by increasing nutritional tolerance.

There is no study in the literature on the effect of abdominal massage on critical patients in pediatric intensive care, and studies are needed in this area.

ELIGIBILITY:
Inclusion criteria: Obtaining parental permission and a signed informed voluntary consent form; the child being aged between 1 and 24 months; receiving mechanical ventilation support for at least 48 hours and being endotracheally intubated; receiving full enteral nutrition during this period; being fed via a nasogastric/orogastric tube and receiving the same type of enteral formula; and receiving sedation.

Exclusion criteria: A high (15%-30%) or very high (>30%) expected mortality rate according to the PRISM III (Pediatric Risk of Mortality) score; planned extubation; lack of anatomical integrity of the gastrointestinal system (history of abdominal surgery, presence of gastrostomy or stoma, presence of tracheostomy); hemodynamic instability; and the presence of severe neurological conditions such as intracranial hemorrhage, increased intracranial pressure, or cranial tumors.

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Variation of gastric residue measurement compared to abdominal massage | Three days
  The gastric residue will be checked by the nurses with a feeding syringe and recorded on the investigation form. Before each feeding, gastric residue will be checked. Before and after the massage results will be compared.
Bowel sounds in minutes / numbers | Three days
  Bowel sounds are listened to with a stethoscope on four quadrants for one minute.
Presence of defecation in terms of days / frequency | Three days
  It is recorded how many times the patient defecation during the day.
Measurement of abdominal circumference in centimeters | Three days
  The abdominal circumference of the patient is measured with the help of a tape measure.
Presence of abdominal distension | Three days
  The abdomen of the patient is examined manually and evaluated in terms of distension.
Presence of vomiting in terms of days / frequency | Three days
  How many times the patient vomited during the day is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Sümeyye Kalaycı, Principal Investigator — Bakırkoy Dr.Sadi Konuk Training and Research Hospital, Pediatric Intensive Care Unit
Locations (1):
- Bakırkoy Dr. Sadi Konuk Training and Research Hospital, Bakırköy, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Badini Pourazar, S., Shirinabadi Farahani, A., Ghahri Sarabi, A., Pourhoseingholi, M. A. ve Dehghan, K. The Effect Of Abdominal Touch On Nutritional Tolerance İn Premature Infants: A Randomized Controlled Clinical Trail. International Journal Of Pediatrics, 2018; 6(8): 8119-8128.
- [Background] Dehghan M, Fatehi Poor A, Mehdipour-Rabori R, Ahmadinejad M. Effect of abdominal massage on prevention of aspiration in intubated and enterally fed patients: A randomized controlled trial. J Complement Integr Med. 2020 Sep 23;17(3). doi: 10.1515/jcim-2017-0124. PMID 31710593
- [Background] Demiray, A, Kuzyaka, İ, Açıl, A, İlaslan, N. Evaluation of Intensive Care Patients with Enteral Nutrition in Terms of Nutrition Process and Possible Complications. Düzce University Institute of Health Sciences Journal. 2020; 10 (3), 289-296. DOI: 10.33631 / duzcesbed.599143
- [Background] Fruhwald S, Holzer P, Metzler H. Intestinal motility disturbances in intensive care patients pathogenesis and clinical impact. Intensive Care Med. 2007 Jan;33(1):36-44. doi: 10.1007/s00134-006-0452-7. Epub 2006 Nov 18. PMID 17115132
- [Background] Ghasemi, M., Najafian, B., Khosravi, M., Nekavand, M. Effect of Abdominal Massage on Gastric Residual Volume and Weight Gain of Premature Infants Admitted in NICU. Canon Journal of Medicine. 2019; 1(2), 49-54. doi: 10.30477/cjm.2019.87285
- [Background] Gürkan A, Gülseven B. ENTERAL NUTRITION: CURRENT APPROACHES TO CARE. Anatolian Journal of Nursing and Health Sciences. 2013; 16 (2): 116-122.
- [Background] Haghshenas Mojaveri, M., Jafarian Amiri, S. R., Dalili, H., Khafri, S. ve Hamed, F. The Effect Of Abdominal Massage On The Feeding Tolerance Of Neonates With Very Low Birth Weight. Iranian Journal Of Pediatrics. 2020; 30(2).
- [Background] Kim HY, Bang KS. The effects of enteral feeding improvement massage on premature infants: A randomised controlled trial. J Clin Nurs. 2018 Jan;27(1-2):92-101. doi: 10.1111/jocn.13850. Epub 2017 Jun 28. PMID 28415135
- [Background] Koçhan, E. And Akın, S. Evaluation of Nurses' Knowledge Level Regarding Enteral and Parenteral Nutrition Practices. J Acad Res Nurs, JAREN. 2018; 4 (1), 1-14.
- [Background] Martinez EE, Bechard LJ, Mehta NM. Nutrition algorithms and bedside nutrient delivery practices in pediatric intensive care units: an international multicenter cohort study. Nutr Clin Pract. 2014 Jun;29(3):360-7. doi: 10.1177/0884533614530762. Epub 2014 Apr 16. PMID 24740498
- [Background] Martinez EE, Douglas K, Nurko S, Mehta NM. Gastric Dysmotility in Critically Ill Children: Pathophysiology, Diagnosis, and Management. Pediatr Crit Care Med. 2015 Nov;16(9):828-36. doi: 10.1097/PCC.0000000000000493. PMID 26218259
- [Background] Momenfar F, Abdi A, Salari N, Soroush A, Hemmatpour B. Studying the effect of abdominal massage on the gastric residual volume in patients hospitalized in intensive care units. J Intensive Care. 2018 Aug 10;6:47. doi: 10.1186/s40560-018-0317-5. eCollection 2018. PMID 30116533
- [Background] Rad, Z. A., Haghshenas, M., Javadian, Y., Hajiahmadi, M., & Kazemian, F. The Effect Of Massage On Weight Gain İn Very Low Birth Weight Neonates. Journal Of Clinical Neonatology. 2016; 5(2), 96.
- [Background] Savran, Y., Limon, M., Tokur, M. E. ve Cömert, B. Factors Associated With Insufficient Nutrition And Effects Of Timely Adequate Nutrition Support On Patient Outcomes İn Intubated Adult Intensive Care Unit Patients. Journal Of Medical And Surgical Intensive Care Medicine. 2016; 7(1), 15-21.
- [Background] Seiiedi-Biarag L, Mirghafourvand M. The effect of massage on feeding intolerance in preterm infants: a systematic review and meta-analysis study. Ital J Pediatr. 2020 Apr 23;46(1):52. doi: 10.1186/s13052-020-0818-4. PMID 32326971
- [Background] Singer P, Blaser AR, Berger MM, Alhazzani W, Calder PC, Casaer MP, Hiesmayr M, Mayer K, Montejo JC, Pichard C, Preiser JC, van Zanten ARH, Oczkowski S, Szczeklik W, Bischoff SC. ESPEN guideline on clinical nutrition in the intensive care unit. Clin Nutr. 2019 Feb;38(1):48-79. doi: 10.1016/j.clnu.2018.08.037. Epub 2018 Sep 29. PMID 30348463
- [Background] Tekin, E., Akan, M., Koca, U., Adıyaman, E., Gökmen, A. N., Özkardeşler, S. and Kılıçaslan, N. Comparison of Different Gastric Residual Volumes in Intensive Care Patients Receiving Enteral Nutrition. Turkish Journal of Intensive Care. 2019; 17 (1), 25-30.
- [Background] Terzi, B., and Kökcü, Ö. D. Different Views on Measuring Gastric Residual Volume in Patients Fed Enterally in the Intensive Care Unit. Journal Of Human Rhythm. 2019; 5 (4), 344-351.
- [Background] Uysal N, Eser I, Akpinar H. The effect of abdominal massage on gastric residual volume: a randomized controlled trial. Gastroenterol Nurs. 2012 Mar-Apr;35(2):117-23. doi: 10.1097/SGA.0b013e31824c235a. PMID 22472671
- [Background] Citak, A., Kalkan, G., Anil, A. B., Agin, H., Akyıldız, B. N., Dursun, O. & Yıldızdas, D. (2018). Pediatric Acute Respiratory Distress Syndrome (PARDS) Protocol. http://cayd.org.tr/files/pediatrik-akut-respiratuar-distres-sendromu-pards-protokolu-0p.pdf